CLINICAL TRIAL: NCT02774057
Title: Randomized Cross-Over Trial of Captafer® vs. Oral Iron Sulfate in the Treatment of Iron Deficiency Anemia in Patients With Inflammatory Bowel Disease
Brief Title: Trial of Captafer® vs. Oral Iron Sulfate in the Treatment of Iron Deficiency Anemia in Patients With IBD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Ala'a Sharara, Professor, Head of Gastroenterology Department, American University of Beirut Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM.AS1.46
Record Dates: First submitted 2016-04-06; First posted 2016-05-17 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Iron Deficiency Anemia; Inflammatory Bowel Disease
Keywords: Captafer®; Iron Sulfate; Iron deficiency anemia; inflammatory bowel disease
MeSH Terms: conditions — Anemia, Iron-Deficiency; Inflammatory Bowel Diseases | interventions — Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Initial therapy with Captafer® (Experimental): This arm will consist of 10 patients who will begin Captafer® therapy twice daily for 6 weeks, then undergo a 2 week washout period before crossing over to Iron Sulfate therapy twice daily for an additional 6 weeks.
  Interventions: Drug: Captafer®; Drug: Iron Sulfate
- Initial therapy with Iron Sulfate (Experimental): This arm will consist of 10 patients who will begin Iron Sulfate therapy twice daily for 6 weeks, then undergo a 2 week washout period before crossing over to Captafer® therapy twice daily for an additional 6 weeks.
  Interventions: Drug: Captafer®; Drug: Iron Sulfate

INTERVENTIONS:
Drug: Captafer® — 2 pills daily. Contains
  * Vitamin C, known for its property to facilitate iron absorption by reducing iron to the reduced ferrous state necessary for uptake;
  * Vitamin E, an antioxidant, along with vitamin C it protects Fe++;
  * Folic acid, necessary to prevent megaloblastic anemia and abnormalities in the fetal nervous system, vital during pregnancy;
  * Zinc and Copper which act in different mitochondrial cytochromes-dependent systems and contribute to the use of iron by the biological systems
Drug: Iron Sulfate — 195 mg Iron supplement
  Other Names: Ironorm

SUMMARY:
Ulcerative colitis (UC) is an inflammatory bowel disease (IBD) characterized by chronic inflammation limited to the mucosal layer of the colon. Anemia is a consistent clinical feature of IBD. It is encountered in one third of IBD patients, and is the most common extraintestinal complication of this disease. Anemia has a significant impact on the quality of life of affected patients. Many patients with IBD frequently complain of chronic fatigue commonly caused by anemia and this may be as debilitating to patients as abdominal pain and diarrhea. Anemia in IBD is multifactorial, but is most commonly the result of iron deficiency anemia (IDA) and rarely due to anemia of chronic disease (ACD). Oral iron supplementation has been used traditionally for the treatment of IDA but studies have shown that it may result in disease exacerbation by increasing oxygen free radicals within the lumen of the gut via the Fenton reaction. A recent study done in University Hospitals Birmingham, United Kingdom, has shown that treatment with oral iron results in failure to control anemia in 2 out of 3 IBD patients, which is in part due to the side effects reported by over half of patients. Captafer is a new iron-free oral preparation that contains a special type of oligosaccharides from fish muscle tissue able to make the intestine absorb 3 to 5 times more iron in comparison to the "meat factor". Moreover, Captafer contains other vitamins and supplements that improve anemia.

DETAILED DESCRIPTION:
Twenty patients from the outpatient department at AUBMC will be enrolled in this open label cross-over trial. Patients with active left sided ulcerative colitis, Crohn's disease or active extensive disease with proven IDA will be enrolled. Study patients will receive the treatment following informed consent and will be followed up regularly by the study coordinator for side effects, compliance and adherence. A blood test for hemoglobin and hematocrit and other biomarkers of iron stores and repletion will be done on all patients at baseline and then after 6 weeks and 12 weeks of therapy. In case patients did not tolerate either treatment, they will be switched to the other treatment after a washout period of 2 weeks.

The objective of this study is to compare the efficacy and safety of Captafer which is an iron-free (one fixed non disclosed dose) food supplement given twice daily, to oral iron therapy given at a dose of 195 mg twice daily for the same period of time in an open label cross-over trial in the treatment of iron deficiency anemia in ulcerative colitis and Crohn's disease patients.

Primary endpoint:

Tolerability

Secondary endpoints

Response to iron repletion as using hemoglobin and hematocrit as surrogates Compliance and adherence (monthly pill count)

The study sample size was calculated based on the primary end points of tolerability with a significance level (α) of 0.05, a Power (1-β) of 0.8 with an expected 90% tolerability and adherence for Captafer vs. 50% for oral iron. At these parameters, and taking a non-inferiority limit of 5%, the sample size was calculated to be 20.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Confirmed diagnosis of ulcerative colitis or Crohn's disease
* Proven iron deficiency anemia (Hb<12, transferrin saturation <20%)
* Active left sided colitis or extensive disease (Mayo Score≥5 or Partial Mayo score ≥4)
* Hemoglobin level > 8 g/dL

Exclusion Criteria:

* Age below 18
* Hemoglobin level < 8 g/dL
* Recently hospitalized for disease flare (within 3 months)
* Hemoglobinopathies (including thalassemia)
* Isolated proctitis
* indeterminate colitis
* Known Liver or kidney disease
* Known Celiac disease
* Small bowel resection
* Use of anticoagulants or aspirin
* Known intolerance to oral iron therapy
* Uninvestigated anemia
* Pregnant or lactating women
* Known hypersensitivity to iron sulfate
* Transfusion within the last 4 weeks
* Erythropoetin within the last 8 weeks
* Rheumatoid Arthritis
* History of menometrorrhagia or frequent epistaxis
* Use of Stomach acid-reducing product (classical antacids, Proton Pump Inhibitors, H2-receptors Inhibitors)
* Gastritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Tolerability to Iron sulfate and Captafer® assessed by the number of patients suffering from treatment related side effects using a Treatment Tolerability Assessment Questionnaire 4 point numerical scale (0,1,2,3). | The change of treatment related side effect frequency between baseline (pre-treatment) and end of treatment periods.
  A 4 point (0,1,2,3) numerical scale will be used to assess the presence and frequency of drug related side effects experienced throughout the study, with scoring done at 4 instances: at baseline prior to initiating the first arm of therapy, at the end of the 6 week treatment period, at baseline after the completion of a 2 week washout period and prior to crossing over, and at the end of the cross over 6 week treatment period. Scores are as follows: 0 = Never, 1 = 2 to 3 times per month, 2 = 2 to 3 times per week, and 3 = daily.

SECONDARY OUTCOMES:
Number of patients responding to therapy by measuring the change in the following laboratory measures Hemoglobin, Hematocrit, Iron, Total Iron Binding Capacity, Ferritin, Transferrin Saturation and c-reactive protein. | The change in hemoglobin, hematocrit, iron, TIBC, ferritin, transferrin saturation and c-reactive protein between baseline (pretreatment), following 6 weeks of first arm of therapy, at baseline post 2 week washout period, and 6 weeks post crossover
  Efficacy will be assessed for Captafer® and iron sulfate treatment at the end of the first 6 weeks before crossing over, and at the end of the next 6 weeks after crossing over.
Number of patients compliant and adherent to treatment intake assessed by paper logged pill counts conducted at 4 different time points. | End of 6 weeks before 2 weeks washout, and end of 6 weeks after 2 weeks of washout
  Number of patients compliant and adherent to treatment intake assessed by paper logged pill counts conducted at baseline prior to treatment initiation, after 6 weeks of first arm of treatment completion, at baseline following a 2 week washout period, and at the end of the 6 weeks of therapy following crossing over.

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut - Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No